CLINICAL TRIAL: NCT02671708
Title: Idarubicin+Busulfan+Cyclophosphamide vs Busulfan+Cyclophosphamide Conditioning Regimen for Intermediate-risk Acute Myeloid Leukemia Undergoing Autologous Hematopoietic Stem Cell Transplantation
Brief Title: IDA+BUCY vs BUCY Conditioning Regimen for Intermediate-risk AML Undergoing Auto-HSCT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Third Affiliated Hospital, Sun Yat-Sen University (Other); Peking University People's Hospital (Other); Zhujiang Hospital (Other); Guangzhou First People's Hospital (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Qifa Liu, Professor, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IDA+BUCY vs BUCY-AML-2016
Record Dates: First submitted 2016-01-30; First posted 2016-02-02 (Estimated); Last update posted 2020-03-03 (Actual); Status verified 2019-03

CONDITIONS: Autologous Hematopoietic Stem Cell Transplantation; Acute Myeloid Leukemia; Conditioning
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Busulfan; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IDA+BUCY (Experimental): For intermediate-risk AML undergoing auto-HSCT，IDA+BUCY conditioning regimen was IDA 15mg/m2/day on days -12 and -10；BU 3.2 mg/kg/day on days -7 and -4；CY 60 mg/kg/day on days -3 and -2.
  Interventions: Drug: Idarubicin（IDA）; Drug: Busulfan (BU); Drug: Cyclophosphamide (CY)
- BUCY (Active Comparator): For intermediate-risk AML undergoing auto-HSCT，BUCY conditioning regimen was BU 3.2 mg/kg/day on days -7 and -4；CY 60 mg/kg/day on days
  -3 and -2.
  Interventions: Drug: Busulfan (BU); Drug: Cyclophosphamide (CY)

INTERVENTIONS:
Drug: Idarubicin（IDA） — Idarubicin was administered at 15mg/m2/day on days -12 and -10.
  Arms: IDA+BUCY
Drug: Busulfan (BU) — Busulfan was administered at 3.2 mg/kg/day on days -7 to -4.
Drug: Cyclophosphamide (CY) — Cyclophosphamide was administered at 60 mg/kg/day on days -3 to -2.

SUMMARY:
Autologous hematopoietic stem cell transplantation (Auto-HSCT) is an effective alternative to allogeneic HSCT for intermediate-risk acute myeloid leukemia (AML) without HLA-matched donors. At present, the best conditioning regimen for AML undergoing auto-HSCT remains in discussion. In this study, the safety and efficacy of IDA+BUCY and BUCY myeloablative conditioning regimens in intermediate-risk AML undergoing auto-HSCT are evaluated.

DETAILED DESCRIPTION:
Auto-HSCT is an effective alternative to allogeneic HSCT for intermediate-risk AML without HLA-matched donors. BUCY conditioning regimen is the standard myeloablative regimen. However, auto-HSCT with BUCY conditioning regimen appears to have higher relapse rate. To reduce the relapse rate, IDA is added in the conditioning regimen. In this study, the safety and efficacy of IDA+BUCY and BUCY myeloablative conditioning regimens in intermediate-risk AML patients undergoing auto-HSCT are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Intermediate-risk AML
* Achieving CR after one cycle induction,then receiving three cycles of consolidation therapy including moderate and high doses of Ara-c combined regimens
* With negative MRD before mobilization and collect of peripheral blood stem cells
* Without HLA-matched donors (related and unrelated)
* Refusal of haploidentical hematopoietic stem cell transplantation

Exclusion Criteria:

* Any abnormality in a vital sign (e.g., heart rate, respiratory rate, or blood pressure)
* Patients with any conditions not suitable for the trial (investigators' decision)

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2016-01; Primary Completion 2019-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
leukemia relapse rate | 2 year

SECONDARY OUTCOMES:
overall survival (OS) | 2 year
disease-free survival (DFS) | 2 year
transplant-related mortality (TRM) | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Liu, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Liu H, Huang F, Zhang Y, Wu M, Xu N, Fan Z, Sun Z, Li X, Lin D, Xiong Y, Liu X, Lin R, Shi P, Xu J, Wang Z, Li X, Sun J, Liu Q, Xuan L. Idarubicin plus BuCy versus BuCy conditioning regimens for intermediate-risk acute myeloid leukemia in first complete remission undergoing auto-HSCT: An open-label, multicenter, randomized phase 3 trial. Am J Hematol. 2023 Mar;98(3):408-412. doi: 10.1002/ajh.26800. Epub 2023 Jan 1. PMID 36588387